CLINICAL TRIAL: NCT05583123
Title: Evaluation of the One-piece Zirconia Abutments and Two-piece Zirconia Abutments With Titanium Bases for Single Implant Crowns in Esthetic Region: a Randomized Split-mouth Clinical Trial With 1-year Follow-up
Brief Title: One-piece and Two-piece Zirconia Abutments in Single Implant Crowns in Esthetic Region
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH9th-20-12
Record Dates: First submitted 2022-03-06; First posted 2022-10-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Partial-edentulism

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPZAs group (OG) (Experimental): one-piece zirconia abutments (OPZAs)
  Interventions: Device: restored abutment (OPZAs)
- TPZAs group (TG) (Active Comparator): two-piece zirconia abutments (TPZAs) with friction-fitted titanium bases
  Interventions: Device: restored abutment (TPZAs)

INTERVENTIONS:
Device: restored abutment (OPZAs) — The restorations will be restored by the OPZAs
  Arms: OPZAs group (OG)
Device: restored abutment (TPZAs) — The restorations will be restored with the TPZAs with friction-fitted titanium bases.
  Arms: TPZAs group (TG)

SUMMARY:
The goal of this clinical trail is to evaluate the clinical, radiological and immunological outcomes of the one-piece zirconia abutments (OPZAs) and two-piece zirconia abutments (TPZAs) with friction-fitted titanium bases in single implant crowns in aesthetic region. The main question it aims to answer is:

whether the mechanical properties of one-piece zirconia abutments are the same as those of two-piece zirconia abutments.

Participants who have two missing teeth in aesthetic region will receive the OPZAs for one restoration and the TPZAs for the other.

Researchers will compare OPZAs group (OG) and TPZAs group (TG) to see the clinical, radiological and immunological outcomes of the two.

DETAILED DESCRIPTION:
Objective: To evaluate the clinical, radiological and immunological outcomes of the one-piece zirconia abutments (OPZAs) and two-piece zirconia abutments (TPZAs) with friction-fitted titanium bases in single implant crowns in aesthetic region.

Materials and methods: The study is a single center, split-mouth and randomized controlled clinical trial. Eligible sites of patients will be randomly assigned into two groups: OPZAs group (OG) and TPZAs group (TG). Survival rates, mechanical complication rates, bleeding on probing (BOP%), probing depth (PD), modified plaque index (mPI), marginal bone loss (MBL), concentrations of pro-inflammatory cytokines (TNF-α, IL-6) in peri-implant crevicular fluid (PICF), and pink esthetics score/white esthetics score (PES/ WES) will be evaluated.

Discussion: Results of the present study will help to evaluate the clinical, radiological and immunological outcomes of OPZAs and TPZAs with friction-fitted titanium bases in single implant crowns in aesthetic region and provide evidence for the effects of two types abutments on the health of peri-implant soft and hard tissue.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18;
2. patients with two missing teeth in esthetic region and plan to be restored with two single implant crowns;
3. adjacent to natural teeth;
4. absence of oral mucosal disease and oral infection;
5. implants with conical connection (Nobel Active, Nobel Biocare® or NobelReplace Conical Connection, Nobel Biocare®);
6. patients with the willingness to participate in the present study.

Exclusion Criteria:

1. heavy smokers (>10 cigarettes/day);
2. uncontrolled periodontitis (Full mouth plaque score>20%, full mouth bleeding score>25%, residual pocket depth>5mm);
3. with systematic diseases that may affect implant therapy, such as uncontrolled diabetes mellitus (Fasting blood-glucose>7.2mmol/L, Glycosylated hemoglobin >7%), current intake of bisphosphonates (treatment for malignancy), pregnant(or plan to get pregnant), with history of radiation therapy in head and neck region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical complications rates | 1 year
  Veneer chipping, abutments or implants fracture, screw loosening or fracture and other mechanical complications will be recorded during the 1-year follow-up.

SECONDARY OUTCOMES:
Survival rates | 1 year
  The survival rate was defined as the percentage of success implants and remained crowns which never been replaced.
Peri-implant conditions-BOP% | 1 year
  peri-implant conditions included bleeding on probing% (BOP%)
Peri-implant conditions-PD | 1 year
  pocket probing depth (PD) in mm
Peri-implant conditions-mPI | 1 year
  modified plaque index (mPI).
Marginal bone loss (MBL) | 1 year
  Peri-apical radiographs with paralleling technique will be performed on the day of final restorations delivery and 1 year later. The implant length is used as calibration reference. The distance between restoration margin and the most coronal level of implant-bone contact will be recorded. The final result calculate as the mean value of mesial and distal sites. The alteration of the distance between baseline and 1-year follow-up is defined as the MBL.
Pro-inflammatory cytokines in peri-implant crevicular fluid (PICF) | 1 year
  We will collect the patients' PICF with the paper strip (PerioPaper Strips; Oraflow Inc., Smithtown, NY, USA) at 1-year follow-up to access differences in pro-inflammatory cytokines (IL-6 and TNF-α) between two groups. Enzyme-linked immunosorbent assay (ELISA) will be used to analyzed PICF and evaluated the concentrations of cytokines. The PICF collection method and cytokines determination referred to Christopher A. Barwacz et al.
PES | 1 year
  In this study, pink aesthetic score (PES) will be applied for the objective esthetic assessment of the final restoration. We will take patients' intraoral photos by the camera (D70, Nikon, Tokyo, Japan) at 1 year follow up. The aesthetic effect will be assessed by two specific dentists independently. They will asked to give scores for variables of PES (Mesial papilla, distal papilla, level of soft-tissue margin, soft-tissue contour, alveolar process and soft-tissue color and texture) and WES (Tooth form, tooth volume/outline, color, surface texture and transparency) with the 0-1-2 scoring system. Final PES/WES is the sum of the two.
WES | 1 year
  In this study, white esthetic score (WES) will be applied for the objective esthetic assessment of the final restoration. We will take patients' intraoral photos by the camera (D70, Nikon, Tokyo, Japan) at 1 year follow up. The aesthetic effect will be assessed by two specific dentists independently. They will asked to give scores for variables of PES (Mesial papilla, distal papilla, level of soft-tissue margin, soft-tissue contour, alveolar process and soft-tissue color and texture) and WES (Tooth form, tooth volume/outline, color, surface texture and transparency) with the 0-1-2 scoring system. Final PES/WES is the sum of the two.

CONTACTS AND LOCATIONS:
Overall Officials: Hongchang Lai, Professor, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- =Shanghai Ninth People's Hospital, China, Shanghai, Shanghao, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05583123/Prot_SAP_000.pdf